CLINICAL TRIAL: NCT02010112
Title: Clinical Validation Study to Evaluate Presence of H. Pylori With 13C-Urea Breath Test Using the Dual Mode BreathID® Hp System Compared to Congruent Biopsy Results
Brief Title: Bag Mode BreathID Hp Validation Versus Endoscopy in Detection of Helicobacter Pylori
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: DM-MPBA-0813
Record Dates: First submitted 2013-12-05; First posted 2013-12-12 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: H.Pylori

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Initial Diagnosis Cohort (Experimental): Subjects with clinical indication of H.pylori infection will undergo breath test compared to routine clinical standard of care- endoscopy
  Interventions: Other: Breath Test Collection bags

INTERVENTIONS:
Other: Breath Test Collection bags — Breath Collection bags will be used to collect breath of subjects before and after ingestion of 13-C breath test substrate
  Other Names: IDKit Two

SUMMARY:
A new method of breath collection for testing for Helicobacter Pylori infection has been developed by Exalenz. In this study, it will be compared to the gold standard- endoscopy results to prove its accuracy.

DETAILED DESCRIPTION:
This study will validate a breath collection method by comparing a newly developed breath test kit, IDkit:Hp™ TWO using breath collection bags, to congruent biopsy results (a composite reference standard by analyzing specimens with microbial culture, histological examination and rapid urease test- RUT) in detecting H.Pylori

ELIGIBILITY:
Inclusion Criteria:

* Present with clinical indication of H. pylori and candidate for upper endoscopy
* Have the ability and willingness to sign the Informed Consent Form for initial diagnosis cohort
* Naive to treatment in the past 18 months
* No known H.pylori status (no conclusive test results within last 6 months)

Exclusion Criteria:

* Participation in other interventional trials
* Antibiotics and/or Bismuth preparations within four (4) weeks prior to breath test
* PPI (proton pump inhibitors) or H2 blockers within two (2) weeks prior to breath test
* Pregnant or breastfeeding women
* Allergy to test substrates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
overall percent agreement | 21 days
  The primary study endpoint is the performance measure (overall percent agreement) in initial diagnosis (presence/ absence of H.pylori) between biopsy results and bag mode breath test.

SECONDARY OUTCOMES:
overall percent agreement | 21 days
  The performance measure (overall percent agreement) in post-therapy diagnosis (presence/ absence of H.pylori) between the Dual Mode BreathID® Hp System when using only one pair of IDkit:Hp™ TWO breath collection bags measured within 9 days and congruent biopsy results

CONTACTS AND LOCATIONS:
Overall Officials: Melina Arazy, M.D., Study Director — VP of clinical affairs, Exalenz
Locations (9):
- United States (9):
  - Digestive Disease Associates, PA, Baltimore, Maryland
  - Metropolitan Gastroenterology Group, Chevy Chase, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Digestive Health Care, Ocean Springs, Mississippi
  - Montefiore Hospital, The Bronx, New York
  - Omega Medical Research, Warwick, Rhode Island
  - Clinical Research Solutions, Jackson, Tennessee
  - JM Research, Houston, Texas
  - Bon Secours Health System, Richmond, Virginia